CLINICAL TRIAL: NCT05613829
Title: Preoperative Frailty Index and 90-day Mortality After a Burn Surgery
Brief Title: Frailty Index and Mortality After a Burn Surgery
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, Professor, Asan Medical Center
Other Study IDs: 2022-006
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Burns; Frailty
MeSH Terms: conditions — Burns; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with burn injury
  Interventions: Other: Burn surgery

INTERVENTIONS:
Other: Burn surgery — Patients underwent burn surgery

SUMMARY:
Frailty is a condition of a reduced physiological reserve and is associated with postoperative morbidity and mortality. We evaluated the impact of preoperative frailty index (CFI) on 90-day mortality after a burn surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with burn injuries were admitted to the burn ICU.

Exclusion Criteria:

* Patients with incomplete medical records were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years who were admitted to the burn ICU from 2012 to 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1118 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality | Postoperative 90 days
  Mortality after burn surgery

CONTACTS AND LOCATIONS:
Overall Officials: Young Joo Seo, Principal Investigator — Hangang Sacred Heart Hospital; Young-Kug Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical Center, Seoul, South Korea